CLINICAL TRIAL: NCT06977087
Title: The Efficacy of Prospective Mental Imagery in Enhancing Approach Motivation Among Socially Anxious Individuals: A Randomized Controlled Trial
Brief Title: The Efficacy of Prospective Mental Imagery in Enhancing Approach Motivation Among Socially Anxious Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Christoph Benke, Principal Investigator, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Trau dich! 2.0
Record Dates: First submitted 2025-04-30; First posted 2025-05-18 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Social Anxiety; Social Phobia
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducation + Prospective Mental-Imagery Task (Experimental): Prospective mental imagery of post-exposure experience
  Interventions: Behavioral: Psychoeducation; Behavioral: Prospective Mental Imagery
- Psychoeducation + Verbal Reasoning Task (Active Comparator): Verbal reasoning of pro and cons of exposure
  Interventions: Behavioral: Psychoeducation; Behavioral: Verbal Reasoning

INTERVENTIONS:
Behavioral: Psychoeducation — Providing information about social anxiety, role of safety and avoidance behaviors in maintaining social anxiety, rationale for exposure to feared social situations
Behavioral: Prospective Mental Imagery — A standard imagination script is recounted in which participants have successfully mastered the socially feared situation
  Arms: Psychoeducation + Prospective Mental-Imagery Task
Behavioral: Verbal Reasoning — Participants are asked to reflect on the pros and cons of facing the socially feared situation
  Arms: Psychoeducation + Verbal Reasoning Task

SUMMARY:
The efficacy of an online intervention aimed at enhancing approach motivation and behavioral engagement in confronting anxiety-inducing social situations is examined among individuals with elevated social anxiety. Participants will receive psychoeducation, followed by either a prospective mental-imagery task or a verbal reasoning task. Efficacy of the intervention is measured by ratings of experienced and anticipated pleasure, approach motivation and self-reported engagement with feared situations one week later.

DETAILED DESCRIPTION:
With numerous studies demonstrating its long-term effectiveness, exposure therapy is currently considered the leading evidence-based treatment for anxiety disorders. However, a major limitation in its application is that patients often discontinue treatment due to their unwillingness to confront themselves with the feared situation. Considering that targeting avoidance behaviors and maladaptive fear responses are at the core of exposure therapy, strategies are needed to enhance both approach motivation as well as behavioral engagement with the feared situation. Among individuals with depression, prospective mental imagery has been demonstrated to increase motivation and behavioral engagement in pleasurable activities by elevating anticipated reward as well as anticipatory and anticipated pleasure ('motivational amplifier' hypothesis). Given alterations in motivational and reward processes in individuals with social anxiety, prospective mental imagery may enhance reward anticipation and facilitate approach motivation and engagement in exposure to socially feared situations. The current online study will compare the use of a prospective mental-imagery task to an active control group (verbal reasoning) in improving approach motivation and behavioral engagement with feared situations in individuals with heightened social anxiety. Participants in both conditions will receive psychoeducation. Participants in the experimental group will vividly imagine themselves successfully mastering the feared social situation. Participants in the control condition are asked to reflect on the pros and cons of confronting themselves with the feared social situation. Approach motivation as well as reward anticipation, anticipated and anticipatory pleasure will be assessed before and after the imagery or verbal reasoning task. Engagement with the feared social situation will be assessed one week later. Aim of the randomized controlled trial is to investigate whether prospective mental imagery is effective in enhancing self-reported motivation and engagement with feared situations compared to an active control group. In an exploratory analysis, we will examine whether the efficacy of the prospective imagery training is modulated by individuals' levels of reward sensitivity and anhedonia.

ELIGIBILITY:
Inclusion Criteria:

* Elevated score on Mini-Social Phobia Inventory (Mini-SPIN) > 6
* Moderate fear and avoidance of two specified social situations (i.e., giving a stranger a compliment and asking for a restaurant recommendation), each rated above 5 on a Likert scale ranging from 0 (not at all) to 10 (extremely), respectively
* Avoidance of the two specified social situations (i.e., giving a stranger a compliment and asking for a restaurant recommendation), indicated by not having engaged in either behaviors in the past 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Anticipatory Pleasure | Baseline (prior to the assigned intervention) and immediately post-intervention (following the prospective mental imagery or verbal reasoning task)
  2-item questionnaire on a scale 0 (not at all) to 100 (extremely) assessing current pleasure when imaging approaching and having approached the feared situations.
Anticipated Pleasure | Baseline (prior to the assigned intervention) and immediately post-intervention (following the prospective mental imagery or verbal reasoning task)
  2-item questionnaire on a scale 0 (not at all) to 100 (extremely) assessing expected pleasure when approaching and having approached the feared situations.
Reward Anticipation | Baseline (prior to the assigned intervention) and immediately post-intervention (following the prospective mental imagery or verbal reasoning task)
  2-item questionnaire on a scale 0 (not at all) to 100 (extremely) assessing expected reward related to approaching and having approached the feared situations.
Motivation | Baseline (prior to the assigned intervention) and immediately post-intervention (following the prospective mental imagery or verbal reasoning task)
  Self-reported motivation to approach the feared situations on a scale of 0 (not at all) to 100 (extremely).
Frequency of Exposure | Post-treatment (i.e., 7 days after baseline)
  Self-reported frequency of exposure to the feared situations.

SECONDARY OUTCOMES:
Social Phobia Inventory (SPIN) | Change from baseline to post-treatment (i.e., 7 days)
  17-item questionnaire on a 5-point Likert scale (0 = 'not at all'; 4 = 'extremely') assessing symptom severity related to social anxiety (i.e., fear, avoidance, physical symptoms). Total range score: 0 to 68. Higher scores indicating greater severity of social anxiety.
Mood State Questionnaire | Baseline (prior to the assigned intervention) and immediately post-intervention (following the prospective mental imagery or verbal reasoning task)
  6-item assessment using a 7-point bipolar Likert scale to measure a person's current mood across three dimensions: energetic arousal, valence, and calmness. Higher scores indicating higher energetic arousal, more positive valence, and greater calmness.
Liebowitz Social Anxiety Scale (LSAS) | Change from baseline to post-treatment (i.e., 7 days)
  24-item questionnaire on a 4-point Likert scale (fear: 0 = 'none'; 3 = 'severe'; avoidance: 0 = 'never'; 3 = 'usually') assessing both fear/anxiety and avoidance of social situations, respectively. Total range score: 0 to 144. Higher scores indicating greater fear and avoidance as well as severity of social anxiety.
Patient Health Questionnaire-9 (PHQ-9) | Baseline
  9-item questionnaire on a 4-point Likert scale (0 = 'not at all'; 3 = 'nearly every day') assessing the presence and severity of depressive symptoms. Total range score: 0 to 27. Higher scores indicating more severe depression.
Positive and Negative Affect Schedule (PANAS) | Baseline
  20-item questionnaire on a 5-point Likert scale (0 = 'not at all'; 4 = 'extremely') assessing the presence and intensity of both positive and negative emotions. Total score range for positive affect (PA) and negative affect (NA), respectively: 0 to 50. Higher scores indicate on either scale indicate a higher level of that emotion.
Snaith-Hamilton-Pleasure-Scale (SHAPS) | Baseline
  14-item questionnaire on a 4-point Likert scale (0 = 'strongly disagree'; 3 = 'strongly agree') measuring anhedonia. Total score range: 0 to 42. Higher total scores indicate greater levels of anhedonia.
Positive Valence System Scale (PVSS-21) | Baseline
  21-item questionnaire on a 9-point Likert scale (1= 'extremely untrue of me'; 9 = 'extremely true of me') assessing an individual's response to various types of rewards in daily life. Total score range: 21 to 105. Higher scores indicating a greater tendency to experience pleasure and respond to rewards.
Vividness of Mental Imagination | Immediately after assigned interventions (prospective mental imagery and verbal reasoning task) at baseline
  Vividness of imagination on a scale from 0 (not at all) to 100 (extremely vivid) assessed immediately after prospective mental-imagery and verbal reasoning task.
Verbal Reasoning | Immediately after assigned interventions (prospective mental imagery and verbal reasoning task) at baseline
  Intensity of reflection on the pros and cons of seeking out the feared situation on a scale from (not intensive at all) to 100 (extremely intensive) assessed after prospective mental-imagery and verbal reasoning task.

CONTACTS AND LOCATIONS:
Locations (1):
- Germany Philipps University, Marburg, Germany

REFERENCES:
- [Background] Hallford DJ, Farrell H, Lynch E. Increasing anticipated and anticipatory pleasure through episodic thinking. Emotion. 2022 Jun;22(4):690-700. doi: 10.1037/emo0000765. Epub 2020 Jun 18. PMID 32551746
- [Background] Renner F, Werthmann J, Paetsch A, Bar HE, Heise M, Bruijniks SJE. Prospective Mental Imagery in Depression: Impact on Reward Processing and Reward-Motivated Behaviour. Clin Psychol Eur. 2021 Jun 18;3(2):e3013. doi: 10.32872/cpe.3013. eCollection 2021 Jun. PMID 36397959
- [Background] Renner F, Murphy FC, Ji JL, Manly T, Holmes EA. Mental imagery as a "motivational amplifier" to promote activities. Behav Res Ther. 2019 Mar;114:51-59. doi: 10.1016/j.brat.2019.02.002. Epub 2019 Feb 5. PMID 30797989
- [Background] Ji JL, Geiles D, Saulsman LM. Mental imagery-based episodic simulation amplifies motivation and behavioural engagement in planned reward activities. Behav Res Ther. 2021 Oct;145:103947. doi: 10.1016/j.brat.2021.103947. Epub 2021 Aug 15. PMID 34433114